CLINICAL TRIAL: NCT05588973
Title: Pilot Double-blind Randomized Controlled Clinical Trial for the Prevention of Radiodermatitis in Breast and Head and Neck Cancer Patients in Cyprus
Brief Title: Prevention of Radiodermatitis in Breast and Head and Neck Cancer Patients in Cyprus
Acronym: MEDISKIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Angelos Kassianos (Other)
Collaborators: German Oncology Center, Cyprus (Other); RSL Revolutionary Labs Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Angelos Kassianos, Lecturer, Cyprus University of Technology
Organization: Cyprus University of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CUT_DN_02; RESTART 2016-2020 SEED (Other Grant/Funding Number: Cyprus Research and Innovation Foundation)
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Cancer; Breast Cancer
Keywords: cancer; breast cancer; quality of life; RCT
MeSH Terms: conditions — Head and Neck Neoplasms; Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: The present study is a double-blinded pilot randomized controlled trial with skin cosmetic products aimed at breast and head and neck cancer patients who will undergo radiation therapy. For the study, individuals will be sought from the German Oncology Center of Limassol. The study will include 80 patients of the German Oncology Center who will be diagnosed with breast cancer and will undergo radiotherapy and 20 patients with head and neck cancer who will also undergo radiotherapy. Individuals included in the study will be over 18 years of age and will have signed written consent to participate in the program. This study will involve 100 patients. Patients will be randomized, (giving a number to each patient) into 2 homogeneous groups of 50 people, either to the control group using panthenol (placebo), or to the intervention group using MEDISKIN.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 50 patients will be randomized to the MEDISKIN group and 50 to the panthenol group. Everyone will start using their cream from the start of the treatment and will continue for 2 weeks after the end of the radiation therapy (twice a day). If there are cases of patients using panthenol and it is deemed necessary based on symptoms to use MEDISKIN then they will automatically change group. Before starting to use the skin cosmetic products, patients will be asked to test the product for any allergic reactions. The "mini-patch test" which is standard of practice is carried out by using the substance on the inner elbow or wrist for 24 hours and observing for any reactions.
  Interventions: Other: MEDISKIN cream
- Control group (Placebo Comparator): The group will be using panthenol istead of the MEDISKIN product
  Interventions: Other: Panthenol cream

INTERVENTIONS:
Other: MEDISKIN cream — MEDISKIN cream with collagen
  Arms: Intervention group
Other: Panthenol cream — Panthenol cream
  Arms: Control group

SUMMARY:
The treatment of cancer as a multidimensional disease has improved in recent years with the development of new chemotherapies, targeted biological therapies or radiation therapy protocols and have led to an overall improvement in the survival of oncology patients. These treatments often cause adverse effects on the skin, which can be accompanied by physical and mental suffering and have a significant impact on patients' quality of life. Improving the quality of life of patients is today a therapeutic challenge. The objective of this clinical study is to assess the tolerability of an innovative skin cosmetic product that will be developed specifically for use during curative anticancer treatments, as well as to study the impact on quality of life of skin side effects caused by the treatments.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age,
* understand and be able to provide signed consent for the purpose of the research,
* be diagnosed with breast or head and neck cancer,
* undergo subfractionated radiotherapy of the breast in 15 sessions of a total dose of 40-42Gy, with or without the administration of a booster dose (boost),
* to know the Greek or English language well
* any wound should have healed after radiotherapy. The criteria will be evaluated by the medical staff of the hospital.

Exclusion Criteria:

* those who do not meet the aforementioned inclusion criteria as well as:
* those who suffer from inflammatory cancer,
* those who have untreated wounds and/or other serious dermatological problems
* those with severe/extensive burns
* those who suffer from serious mental disorders (dementia, drug addiction, etc.) that require intensive treatment or monitoring,
* those who have a sensitivity/allergy to any of the product's ingredients. The criteria will be evaluated by the medical staff of the hospital.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Dermatological Quality of Life | Baseline (1 month before radiotherapy), during therapy (15 days), 1 week post therapy, 1 month later
  Questionnaire SKINDEX-17 | The Skindex-17 is a dermatological HRQoL instrument that was derived from the Skindex-29 using Rasch psychometric analysis. It consists of 17 items instead of 29, and answers are given on a four-point scale instead of a five-point scale. The tool offers 2 measures: psychosocial health and symptomatology with higher scores reporting increased quality of life and symptomatology respectively. Change in dermatological quality of life immediately after treatment will be used as the primary outcome.

SECONDARY OUTCOMES:
Dermatological Quality of Life (b) | Baseline (1 month before radiotherapy), First day of therapy with Mediskin products (and after radiotherapy), During therapy (15 days), 1 week post therapy
  Dermatology Quality of Life Index Questionnaire | The Dermatological Quality of Life Index (DLQI) is a tool often used by dermatologists to assess the impact of skin disease on quality of life in areas such as work and social activities, as well as patients' symptoms and feelings about their pathological condition. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more the quality of life is reduced/affected. DLQI can also be expressed as a percentage of the maximum possible score of 30 (ie % of 30). There will be 3 measurements during treatment one every 5 days.
Health Related Quality of Life | Baseline (1 month before radiotherapy), First day of therapy with Mediskin products (and after radiotherapy), during therapy (15 days), 1 week post therapy, 1 month later
  EORTC QLQ-C30 Questionnaire | European Organization for Research and Treatment of Cancer Questionnaire that assesses the quality of life of cancer patients (EORTC QLQ - C30) (Aaronson et al 1993, Osaba et al 1994). We will use the validated Greek version of this result version 3. The questionnaire is summed through a specific algorithm into 4 categories: physical function, psychological function, social function and a series of symptoms such as pain, fatigue, etc. A higher score in each means better functioning (in functioning subpscales), better quality of life (in the global quality of life subscale) and worse symptoms (in symptomatology sub-scales). The change in measurement will be used both with the end of treatment as well as 1 month later.
Real time quality of life | During therapy (15 days)
  To better understand the patient's condition during the treatment we will use a mobile application (PRICE EMA app) which was created by researchers of the University of Cyprus, Cyprus University of Technology and CYENS with the data stored in a GDPR compliant cloud based system accessible only through codes and encoded to match the redcap data. We will measure quality of life using an adapted version of the EORTC QLQ C30 global quality of life subscale with a higher score on a 0-100 scale indicating better quality of life, through brief self-reports that patients will complete through in-app notifications. The development of the PRICE methodology and tool is explained here: https://dl.acm.org/doi/abs/10.1145/3491101.3503562?casa_token=_pSlJoCNphIAAAAA:RMI4xGtq2J-T9BJHqDjAU3R-pVx3OdqR0gIRAvNLBHuP6c8gt3YRRO4CryevCopqBOVAZQ-X7_7
Real time anxiety | During therapy (15 days)
  To better understand the patient's condition during the treatment we will use a mobile application (PRICE EMA app) which was created by researchers of the University of Cyprus, Cyprus University of Technology and CYENS with the data stored in a GDPR compliant cloud based system accessible only through codes and encoded to match the redcap data. We will measure anxiety through brief self-reports that patients will complete through in-app notifications using an adapted version of the anxiety sub scale of Hospital Anxiety and Depression Scale (HADS) with higher scores on a 0-21 score indicating higher levels of anxiety symptoms. The development of the PRICE methodology and tool is explained here: https://dl.acm.org/doi/abs/10.1145/3491101.3503562?casa_token=_pSlJoCNphIAAAAA:RMI4xGtq2J-T9BJHqDjAU3R-pVx3OdqR0gIRAvNLBHuP6c8gt3YRRO4CryevCopqBOVAZQ-X7_7
Real time depression | During therapy (15 days)
  To better understand the patient's condition during the treatment we will use a mobile application (PRICE EMA app) which was created by researchers of the University of Cyprus, Cyprus University of Technology and CYENS with the data stored in a GDPR compliant cloud based system accessible only through codes and encoded to match the redcap data. We will measure depression through brief self-reports that patients will complete through in-app notifications using an adapted version of HADS with higher scores on a 0-21 score indicating worse depression symptomatology. The development of the PRICE methodology and tool is explained here: https://dl.acm.org/doi/abs/10.1145/3491101.3503562?casa_token=_pSlJoCNphIAAAAA:RMI4xGtq2J-T9BJHqDjAU3R-pVx3OdqR0gIRAvNLBHuP6c8gt3YRRO4CryevCopqBOVAZQ-X7_7
Real time pain | During therapy (15 days)
  To better understand the patient's condition during the treatment we will use a mobile application (PRICE EMA app) which was created by researchers of the University of Cyprus, Cyprus University of Technology and CYENS with the data stored in a GDPR compliant cloud based system accessible only through codes and encoded to match the redcap data. We will measure pain/irritation through brief self-reports developed for this study that patients will complete through in-app notifications with a higher score on a 0-10 score indicating worse pain symptoms. The development of the PRICE methodology and tool is explained here: https://dl.acm.org/doi/abs/10.1145/3491101.3503562?casa_token=_pSlJoCNphIAAAAA:RMI4xGtq2J-T9BJHqDjAU3R-pVx3OdqR0gIRAvNLBHuP6c8gt3YRRO4CryevCopqBOVAZQ-X7_7
Real time fatigue | During therapy (15 days)
  To better understand the patient's condition during the treatment we will use a mobile application (PRICE EMA app) which was created by researchers of the University of Cyprus, Cyprus University of Technology and CYENS with the data stored in a GDPR compliant cloud based system accessible only through codes and encoded to match the redcap data. We will measure fatigue through brief self-reports developed for this study that patients will complete through in-app notifications with a higher score on a 0-10 score indicating worse fatigue symptoms. The development of the PRICE methodology and tool is explained here: https://dl.acm.org/doi/abs/10.1145/3491101.3503562?casa_token=_pSlJoCNphIAAAAA:RMI4xGtq2J-T9BJHqDjAU3R-pVx3OdqR0gIRAvNLBHuP6c8gt3YRRO4CryevCopqBOVAZQ-X7_7
Socio-demographic questionnaire | Baseline (1 month before radiotherapy)
  Developed for this study
Acceptability questionnaire | First day of therapy with Mediskin products (and after radiotherapy), 1 week post therapy, 1 month post baseline
  Developed for this study with responses in open ended questions that will be analysed descriptively and thematically.

CONTACTS AND LOCATIONS:
Overall Officials: Angelos P. Kassianos, PhD, Study Chair — Cyprus University of Technology
Locations (1):
- Cyprus University of Technology, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided